CLINICAL TRIAL: NCT00024466
Title: Vaccination In Peripheral Stem Cell Transplant Setting For Multiple Myeloma: The Use Of Autologous Tumor Cells/An Allo PSCT
Brief Title: Chemotherapy, Vaccine Therapy, and Stem Cell Transplantation in Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0115; P30CA006973 (NIH); 01-01-17-06 (Other: JHMIRB)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — FANG vaccine; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Experimental): Participants are vaccinated with GVAX one month or more after finishing induction therapy (which is given as per standard of care). Two weeks later, participants go through leukapheresis on protocol, then receive autologous transplant as per standard of care. GVAX is administered eight subsequent times after the autologous transplant.
  Interventions: Biological: GVAX; Procedure: Autologous transplant

INTERVENTIONS:
Biological: GVAX
  Other Names: Autologous tumor vaccine
Procedure: Autologous transplant
  Other Names: Auto BMT; Auto SCT

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Vaccines made from a person's cancer cells may make the body build an immune response to kill cancer cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy. Combining chemotherapy with vaccine therapy and peripheral stem cell transplantation may be effective in treating multiple myeloma.

PURPOSE: Phase I/II trial to study the effectiveness of chemotherapy followed by vaccine therapy and peripheral stem cell transplantation in treating patients who have newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of induction chemotherapy followed by autologous tumor cell vaccine and autologous peripheral blood stem cell transplantation in patients with multiple myeloma.
* Determine the safety of this regimen in these patients.

OUTLINE: Autologous tumor cells are harvested. The vaccine is prepared in vitro by mixing autologous tumor cells with a bystander cell expressing sargramostim (GM-CSF). Patients receive induction chemotherapy followed by autologous tumor cell vaccination (ATCV) once. Patients then undergo autologous peripheral blood stem cell transplantation. At 6 weeks after transplantation, patients receive additional ATCVs every 3 weeks for a total of 8 vaccinations.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA

Initial Presentation

* Age between 18 and 70 years
* ECOG 0 - 2
* Patients with histologically confirmed multiple myeloma with ≥ 30% bone
* marrow involvement and a de novo presentation. One cycle of prior
* chemotherapy for myeloma is allowed. Local radiation therapy is permitted
* Ability to give informed consent
* No existing secondary malignancies and no history of secondary malignancies in the past 5 years (other than a history of carcinoma in situ of the cervix, superficial skin cancer, or superficial bladder cancer)
* No active autoimmune disease, nor a history of any autoimmune disease requiring medical treatment with systemic immunosuppressants
* No corticosteroids within 28 days of tumor harvest
* No major active medical or psychosocial problems that could be exacerbated or complicated by this treatment
* Not pregnant
* HIV negative
* AST/ALT, total bilirubin < threefold normal
* Absolute neutrophil count >500/mm3
* Platelet count >30,000/mm3

Prior to Transplantation

* ECOG performance status of 0 - 2.
* No active/uncontrolled infection.
* Absolute neutrophil count (ANC) >1000/mm3.
* Platelet count >50,000/mm3.
* Hemoglobin >8g/dL
* AST/ALT, total bilirubin <3-fold normal.
* 50% or greater reduction in tumor burden with prior chemotherapy
* Patient has received a minimum of 2 cycles of an accepted induction
* chemotherapy regimen
* Patient fulfills the requirements for standard peripheral stem cell transplantation Prior to Posttransplant Vaccination
* No active/uncontrolled infection
* Absolute neutrophil count (ANC) >1000/mm3
* Platelet count >50,000/mm3
* Hemoglobin >8g/dL
* AST/ALT, total bilirubin <3-fold normal
* No unresolved Grade 3 or 4 adverse events related to the transplant

EXCLUSION CRITERIA

• Failure of autologous tumor-cell processing for vaccine production

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2001-04 (Actual); Primary Completion 2004-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Tumor-specific immune response | Up to 1 year
  Percentage of participants who had a delayed-type hypersensitivity reaction with induration greater than or equal to 5 millimeters to an intradermal injection of irradiated autologous tumor cells.

SECONDARY OUTCOMES:
Grade 3-4 toxicity | Up to 1 year
  Percentage of participants with grade 3-4 toxicity as measured by Common Terminology Criteria for Adverse Events (CTCAE 2.0).

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Borrello, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No